CLINICAL TRIAL: NCT06692439
Title: Acute Heart Failure in Elderly Patients Admitted to the Emergency Department with Acute Dyspnea: a Multimarker Approach Prognostic Study
Acronym: READ-MA-PRONO
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/725
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Acute Heart Failure (AHF); Dyspnoea
Keywords: acute heart failure; dyspnea; prognosis; biomarkers
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- acute heart failure: The presence or absence of acute left heart failure (gold standard) was determined through diagnosis by two experts (a cardiologist and an emergency physician) based on:
  1. Data collected in the ED and during hospitalization: Clinical examination and history, Current medications, Hemodynamic parameters, ECG, Chest X-ray, Emergency interventions, Clinical and paraclinical findings during hospitalization
  2. Biological assays (excluding NT-proBNP)
  3. Echocardiography performed by a cardiologist within 24 hours of admission, including: Left Ventricular Ejection Fraction, Segmental wall motion, Presence of valvular disease, Transmitral flow, Tissue Doppler E' velocity
  anticipated, n = 185/450 (41%)
- no acute heart failure: The presence or absence of acute left heart failure (gold standard) was determined through diagnosis by two experts (a cardiologist and an emergency physician) based on:
  1. Data collected in the ED and during hospitalization: Clinical examination and history, Current medications, Hemodynamic parameters, ECG, Chest X-ray, Emergency interventions, Clinical and paraclinical findings during hospitalization
  2. Biological assays (excluding NT-proBNP)
  3. Echocardiography performed by a cardiologist within 24 hours of admission, including: Left Ventricular Ejection Fraction, Segmental wall motion, Presence of valvular disease, Transmitral flow, Tissue Doppler E' velocity
  anticipated, n = 265/450 (59%)

SUMMARY:
Background and Rationale:

Acute dyspnea is a frequent presenting symptom in emergency departments (ED), with acute heart failure (AHF) being the most common cause leading to hospitalization in elderly patients. AHF in this population presents unique challenges in diagnosis, management, and risk stratification. Current tools for severity assessment and risk stratification (NT-proBNP and echocardiography) have shown limited evolution over the past 20 years and remain insufficient, particularly for elderly patients who predominantly present with heart failure with preserved ejection fraction (HFpEF). Recent European Society of Cardiology (ESC) and American Heart Association (AHA) guidelines specifically call for research on biomarkers within a multi-marker strategy for AHF risk stratification.

Research Hypothesis:

The study hypothesizes that a combination of biomarkers (NT-proBNP, High-sensitivity Troponin I, ST2, Galectin-3, CD146 and suPAR) will provide prognostic value and effectively stratify risk for early outcomes (90-day mortality and hospital readmission) in patients aged ≥75 years presenting to the ED with acute dyspnea and diagnosed with AHF.

Primary Objective:

To evaluate the prognostic value of six biomarkers, both individually and in combination, for predicting 90-day all-cause mortality or ED readmission in elderly patients (≥75 years) presenting with acute dyspnea and diagnosed with AHF.

Study Design:

This is a prospective prognostic study including patients from 7 emergency departments from university and non-university hospitals in France.

Study Population:

(I) Patients aged ≥75 years presenting to the ED with acute dyspnea meeting at least two criteria:

* Respiratory rate ≥25/min
* PaO2 ≤70 mmHg
* SpO2 ≤92% on room air
* PaCO2 ≥45 mmHg and pH ≤7.35
* Oxygen requirement

(ii) Have confirmed AHF diagnosis by two expert reviewers based on clinical data, laboratory results (excluding NT-proBNP), ECG, imaging, and specialized cardiac echo

Primary Endpoint:

Composite endpoint of 90-day all-cause mortality or ED readmission, as recommended by the ESC for evaluating early outcomes in AHF patients.

Analysis plan includes:

* ROC curves for optimal biomarker thresholds
* Kaplan-Meier survival analysis with log-rank tests
* Univariate and multivariate Cox regression analyses
* Bootstrap methods for confidence intervals

ELIGIBILITY:
Inclusion Criteria: Patients aged ≥75 years from the READ cohort (NCT04240067) who:

1. Present to the ED with acute dyspnea meeting at least two criteria:

   * Respiratory rate ≥25/min
   * PaO2 ≤70 mmHg
   * SpO2 ≤92% on room air
   * PaCO2 ≥45 mmHg and pH ≤7.35
   * Oxygen requirement
2. Have confirmed AHF diagnosis by two expert reviewers based on clinical data, laboratory results (excluding NT-proBNP), ECG, imaging, and specialized cardiac echo
3. Provided written consent for data use in the READ-MA-PRONO study

Exclusion Criteria:

* No written consent for data use in the READ-MA-PRONO study

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients aged ≥75 years admitted to the ED for acute dyspnea
Sampling Method: Probability Sample
Enrollment: 185 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of 90-day all-cause mortality or ED readmission, as recommended by the ESC for evaluating early outcomes in AHF patients. | 90-day

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric MAUNY, MD, PhD, Study Chair — CHU Besançon; Marc PUYRAVEAU, MSc, Study Chair — CHU Besançon

IPD SHARING:
Plan to Share IPD: Undecided